CLINICAL TRIAL: NCT07139158
Title: Quadriceps Muscle Oxygenation During Different Lower Limb Tasks in Patients With Patellofemoral Pain: A Cross-Sectional Study
Brief Title: Muscle Oxygenation in Patellofemoral Pain
Status: Completed | Type: Observational
Sponsor: Ankara Medipol University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Selcan Suicmez, Research Assistant, Ankara Medipol University
Other Study IDs: GaziU-FTR-SS-03
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: Patellofemoral Pain, PFP
Keywords: patellofemoral pain; near-infrared spectroscopy; lower extremity; kinesiophobia; physical activity
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Kinesiophobia; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patellofemoral Pain Group
- Pain-free Control Group

SUMMARY:
Patellofemoral joint problems account for a significant portion of knee pain and disability. Among these problems, patellofemoral pain is not directly related to any obvious structural abnormality and is characterized by pain in the retro- or peri-patellar region, particularly during activities such as squatting, running, and climbing stairs. It is commonly seen in the general population. The current literature highlights the tendency of patellofemoral pain to recur and become chronic despite all treatments. Individuals with patellofemoral pain often experience disorders in the neuromuscular function of the quadriceps femoris muscle, which is necessary for knee function and dynamic stability and is frequently suggested to play an important role in the pathophysiology of the disease. A decrease in the tissue's ability to utilize oxygen during exercise or physical activity may lead to permanent dysfunction of the quadriceps femoris muscle. However, no studies have been found in the literature examining changes in oxygenation of the quadriceps femoris muscle in individuals with patellofemoral pain. Therefore, the aim of this study is to investigate changes in oxygenation of the quadriceps femoris muscle in individuals with patellofemoral pain during various exercises and physical activities by comparing them with pain-free individuals.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age
* pain around or behind the patella, which is aggravated by at least one activity that loads the patellofemoral joint during weight bearing on a flexed knee (e.g., squatting, stair ambulation, jogging/running, hopping/jumping)
* the pain persist for at least four months, and be rated at ≥ 3/10 on the Numeric Pain Rating Scale (NPRS)
* vastus medialis muscle adipose tissue thickness <20 mm

Pain-free controls were age- and gender-matched, with vastus medialis muscle adipose tissue thickness <20 mm.

Exclusion Criteria:

* a history of joint surgery
* meniscal and/or ligament injuries
* patellar instability, congenital patellar subluxation/dislocation
* any cardiovascular, congenital, or musculoskeletal disorders that could interfere with the assessment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty-one patients with patellofemoral pain and 20 pain-free controls will be conducted at Ankara Medipol University, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Muscle Oxygenation | Day 1
  Vastus medialis muscle oxygenation will be evaluated with Near-Infrared Spectroscopy at rest, during and after activity.

SECONDARY OUTCOMES:
Kujala Patellofemoral Score Scale | Day 1
  Kujala patellofemoral scoring is a tool that allows functional evaluation of knee complaints related to the patellofemoral structure. Different scoring systems have been developed for knee-specific symptoms; however, only a few of these are focused on patellofemoral pain.The Kujala Patellofemoral Score Scale is graded on a scale of 0 to 100, with 100 being the highest possible score.
International Physical Activity Questionnaire (IPAQ) | Day 1
  Provides information on time spent walking, moderate and vigorous activities, and time spent sitting. Calculation of the total score of the short form includes the sum of the duration (minutes) and frequency (days) of walking, moderate-intensity activity, and vigorous activity. The energy required for activities is calculated with the metabolic equivalent(MET) -minute score. Standard metabolic equivalent (MET) values have been established for these activities.
Adipose tissue thickness | Day 1
  The skinfold thickness of vastus medialis muscle was evaluated with a Skinfold Caliper. Adipose tissue thickness was obtained by dividing the skinfold thickness by two.
Numeric Pain Rating Scale | Day 1
  Numeric pain rating scale is a scale used to quantify pain intensity. It is divided into eleven equal parts; for example 0 - 10. O means that there is no pain at all, 1 - 3 divisional range falls in the mild category pain , 4 - 6 indicates the symptoms of moderate pain while 7 - 10 reading symptoms the severity of pain.
Tampa Kinesiophobia Scale | Day 1
  The Tampa Kinesiophobia Scale is a 17-question questionnaire that assesses avoidance of injury and fear of movement. The scale is scored using a Likert scale (1 = Strongly disagree, 4 = Strongly agree). Items 4, 8, 12 and 16 are reversed to calculate the total score of the scale. The total score is between 17 and 68. As the score of the person increases, it is understood that their kinesiophobia is high. A total score higher than 37 is considered as high kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No